CLINICAL TRIAL: NCT01234259
Title: Evaluation of Safety and Efficacy of Using Venus Freeze™ (MP)2 V2 System for Wrinkles Rhytides and Cellulite Treatment - a Pilot Study
Brief Title: Evaluation of Safety and Efficacy of Using Venus Freeze™ (MP)2 V2 System for Wrinkles Rhytides and Cellulite Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VN-WR- 01
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Wrinkled Structure; Circumference Reduction
Keywords: Wrinkles; rhytides; Cellulite; circumference reduction
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Device: Venus Freeze (MP)2 V2 system
  Interventions: Device: Venus Freeze (MP2 V2 System
- control group: (Sham Comparator): Sham comparator
  Interventions: Device: Venus Freeze (MP2 V2 System

INTERVENTIONS:
Device: Venus Freeze (MP2 V2 System — Facial wrinkles and temporary cellulite and circumference reduction treatments

SUMMARY:
Skin aging is a multifactorial process involving the 3 layers of the skin: Epidermis, dermis and hypodermis.

Radio-frequency (RF) devices have been used for many years for a variety of surgical applications. The energy delivery systems of these established monopolar devices used a 'conductive coupling' delivery system in which energy is concentrated at the periphery of the electrode.

Venus Concept has developed the Venus Freeze (MP)2 V2 system for wrinkles, rhytides and temporary cellulite and circumference reduction treatments. While treating wrinkles rhytides and cellulite, the treatments creates enough thermal effect to induce collagen remodeling with no ablative thermal damage in the epidermis or dermis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females age 30 and up
* Subjects with Fitzpatrick 4 to 9 degrees of elastosis
* Subject able to comprehend and give informed consent for participation in this study
* Subject must commit to all treatments and follow-up visits
* Subject must sign the Informed Consent Form

Exclusion Criteria:

* Subjects with implanted pacemakers, arrhythmias or any other severe known heart disorder
* Subjects with any implantable metal device in the treatment area
* Subjects on any medication that would affect the characteristic of the skin (medical or hormonal), such as "Accutane", within the past 6 months or photosensitizing medications
* Subjects that have had any other invasive or non invasive method of skin therapy or hair removal performed in the past 9 months (in the treated area) Subjects who are scheduled or planned for any other invasive or non invasive method of skin therapy or hair removal in the treated area at the period of the study
* Subjects who have any form of malignant skin cancer on the treatment area
* Subjects with history of keloid formations or hypertrophic scarring
* Pregnant or lactating Subjects
* Subjects with Epilepsy or severe migraines
* Subjects with permanent makeup/ tattoo/ body piercing (in the treated area)
* Subjects with any Infection / abscess / dermatitis/ pains in treatment target area.
* Subjects who suffer from autoimmune disorders or diabetes
* Subjects with clotting disorders
* Subjects are suffering from psychiatric disorders and treated with psychiatric medications.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol
* Concurrent participation in any other clinical study
* Physician objection

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the Venus system for wrinkles rhytides and temporary cellulite and circumference reduction treatment. Efficacy evaluation will include RF, Magnetic Pulse Field and vacuum technology. | 5 months
  Efficacy will be established by skin improvement as a result of the treatment by validated scales. Results will be compared to control group results. The pre - and post-treatment photographs will be compared and assessed by three independent dermatologists.

SECONDARY OUTCOMES:
To evaluate the safety of the Venus Freeze (MP)2 V2 system for wrinkles, rhytides, temporary cellulite and circumference reduction. Safety evaluation will include RF, Magnetic Pulse Field and vacuum technology. | 5 months
  Safety parameters will include adverse events (signs of pain; edema; burn; localized infection; skin pigmentation & texture alterations) occurring as a direct result of the treatment and complaints up to last follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Sprecher, Prof., Principal Investigator — Tel-Aviv Sourasky medical Centre, Israel
Locations (1):
- Sourasky medical Centre, Tel Aviv, Israel